CLINICAL TRIAL: NCT02438410
Title: Correlation of Infliximab Levels With Outcomes in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Darrell S. Pardi, M.D., PI, Mayo Clinic
Other Study IDs: 14-005723
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Results first posted 2022-03-03 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Disease; IBD
Keywords: infliximab; remicade; IBD; Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool and blood laboratory data such as CBC with differential, creatinine, TNF levels, albumin, fecal calprotectin, ESR, CRP, infliximab and antibodies to infliximab levels will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess if infliximab drug levels in subjects with Ulcerative Colitis predict risk of colectomy rate. Additionally, the investigators will estimate an optimal day 4 infliximab level based on the study results.

DETAILED DESCRIPTION:
Infliximab is approved for induction and maintenance of clinical remission and mucosal healing in patients with moderate to severe active ulcerative colitis, in those who have an inadequate response to conventional therapy such as IV steroids. It is typically dosed at 5 mg/kg at 0, 2, and 6 weeks, followed by 5 mg/kg every 8 weeks thereafter. The alternative to rescue medical therapy with infliximab is proctocolectomy with ileal pouch anastomosis, which carries risks including pouchitis, fecal incontinence, pouch failure requiring further surgical procedures and female infertility, or proctocolectomy with permanent end-ileostomy, which many patients wish to avoid. The induction regimen of 3 doses of Infliximab followed by a maintenance dose every 8 weeks is used to achieve response in hopes of avoiding colectomy. Unfortunately, a large proportion of patients are unable to achieve or sustain a clinical response over time and end up getting a colectomy.

Potential implicated pathways in non-responders include fecal wasting of infliximab and factors that accelerate drug clearance such as a large TNF (tumor necrosis factor) or CRP (C reactive protein) burden, anti-infliximab antibodies (ATI), low serum albumin, male sex and larger body size. Patients with severe ulcerative colitis who fail corticosteroids and standard dosing with infliximab usually proceed to proctocolectomy. Optimizing early infliximab blood levels in patients with moderate-severe ulcerative colitis by administering the second dose of infliximab before week 2 could improve the efficacy and further reduce the need for colectomy. However, there is a paucity in the literature as this is a relatively new school of thought. Our study will address this deficit by evaluating the relationship between early drug levels of infliximab in ulcerative colitis and colectomy rates at one and three months.

ELIGIBILITY:
Inclusion Criteria

1. Adults, ages 18-65 years
2. Hospitalized, with a moderate -severe flare. Based on the Mayo Scoring System for Assessment of Ulcerative Colitis Activity (Mayo score of equal or greater than 6)
3. Treatment naïve to anti TNF agents
4. Initiation of infliximab, with or without immunomodulator such as azathioprine
5. Ongoing use of immunomodulators such as azathioprine or 6MP is acceptable. Their initiation or continuation remains at the discretion of the treating physician

Exclusion Criteria

1. Ongoing or prior treatment with Infliximab or other anti TNF agents
2. Ongoing or recent (with in 1 month) administration of rescue cyclosporine
3. Fulminant colitis requiring emergent surgery or toxic megacolon
4. Pregnancy
5. Infectious colitis, for example Clostridium difficile or CMV (cytomegalovirus) colitis
6. Active infection or abscess
7. Untreated latent or active tuberculosis (TB). Those with latent TB who are currently undergoing treatment can be included. Please refer to appendix 1 for more information on specific inclusion and exclusion criteria related to TB testing. Refer to 1.4.2 of appendix 1 for TB screening questions
8. Active malignancy
9. Active or history of Congestive Heart failure (CHF) or those who have received treatment for CHF
10. Active or history of Multiple Sclerosis (MS), or those who have received treatment for MS
11. Prisoners, institutionalized individuals, and individuals who are not capable of giving informed consent
12. Judgement of investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be scheduled to receive clinically indicated infliximab at the discretion of their treating physician during an acute hospitalization with a flare of moderate to severe UC. These will be inpatients at Mayo Clinic Rochester campus or be admitted in Mayo Clinic Health Systems. Endoscopic findings will be noted and those deemed to have moderate to severe disease activity based on the Mayo Scoring System for Assessment of Ulcerative Colitis Activity will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-05; Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell S Pardi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363
- [Background] Molodecky NA, Kaplan GG. Environmental risk factors for inflammatory bowel disease. Gastroenterol Hepatol (N Y). 2010 May;6(5):339-46. PMID 20567592
- [Background] Danese S, Fiocchi C. Ulcerative colitis. N Engl J Med. 2011 Nov 3;365(18):1713-25. doi: 10.1056/NEJMra1102942. No abstract available. PMID 22047562
- [Background] Kornbluth A, Sachar DB; Practice Parameters Committee of the American College of Gastroenterology. Ulcerative colitis practice guidelines in adults (update): American College of Gastroenterology, Practice Parameters Committee. Am J Gastroenterol. 2004 Jul;99(7):1371-85. doi: 10.1111/j.1572-0241.2004.40036.x. PMID 15233681
- [Background] Campbell S, Travis S, Jewell D. Ciclosporin use in acute ulcerative colitis: a long-term experience. Eur J Gastroenterol Hepatol. 2005 Jan;17(1):79-84. doi: 10.1097/00042737-200501000-00016. PMID 15647646
- [Background] Sandborn WJ. A critical review of cyclosporine therapy in inflammatory bowel disease. Inflammatory Bowel Diseases 1995;1:48-63.
- [Background] Jarnerot G, Hertervig E, Friis-Liby I, Blomquist L, Karlen P, Granno C, Vilien M, Strom M, Danielsson A, Verbaan H, Hellstrom PM, Magnuson A, Curman B. Infliximab as rescue therapy in severe to moderately severe ulcerative colitis: a randomized, placebo-controlled study. Gastroenterology. 2005 Jun;128(7):1805-11. doi: 10.1053/j.gastro.2005.03.003. PMID 15940615
- [Background] Waljee A, Waljee J, Morris AM, Higgins PD. Threefold increased risk of infertility: a meta-analysis of infertility after ileal pouch anal anastomosis in ulcerative colitis. Gut. 2006 Nov;55(11):1575-80. doi: 10.1136/gut.2005.090316. Epub 2006 Jun 13. PMID 16772310
- [Background] Penna C, Dozois R, Tremaine W, Sandborn W, LaRusso N, Schleck C, Ilstrup D. Pouchitis after ileal pouch-anal anastomosis for ulcerative colitis occurs with increased frequency in patients with associated primary sclerosing cholangitis. Gut. 1996 Feb;38(2):234-9. doi: 10.1136/gut.38.2.234. PMID 8801203
- [Background] Hahnloser D, Pemberton JH, Wolff BG, Larson DR, Crownhart BS, Dozois RR. The effect of ageing on function and quality of life in ileal pouch patients: a single cohort experience of 409 patients with chronic ulcerative colitis. Ann Surg. 2004 Oct;240(4):615-21; discussion 621-3. doi: 10.1097/01.sla.0000141157.32234.9d. PMID 15383789
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Peyrin-Biroulet L, Deltenre P, de Suray N, Branche J, Sandborn WJ, Colombel JF. Efficacy and safety of tumor necrosis factor antagonists in Crohn's disease: meta-analysis of placebo-controlled trials. Clin Gastroenterol Hepatol. 2008 Jun;6(6):644-53. doi: 10.1016/j.cgh.2008.03.014. PMID 18550004
- [Background] Brandse J.F. MWM, de Bruyn J., Wolbink GJ., Lowenberg M., Ponsioen C., van den Brink G.R., D'Haens G.R. Fecal Loss of Infliximab As a Cause of Lack of Response in Severe Inflammatory Bowel Disease. Gastroenterology May 2013;144:S-36.
- [Background] Ordas I, Mould DR, Feagan BG, Sandborn WJ. Anti-TNF monoclonal antibodies in inflammatory bowel disease: pharmacokinetics-based dosing paradigms. Clin Pharmacol Ther. 2012 Apr;91(4):635-46. doi: 10.1038/clpt.2011.328. Epub 2012 Feb 22. PMID 22357456
- [Background] Gibson DJ, Heetun ZS, Redmond CE, Nanda KS, Keegan D, Byrne K, Mulcahy HE, Cullen G, Doherty GA. An accelerated infliximab induction regimen reduces the need for early colectomy in patients with acute severe ulcerative colitis. Clin Gastroenterol Hepatol. 2015 Feb;13(2):330-335.e1. doi: 10.1016/j.cgh.2014.07.041. Epub 2014 Jul 30. PMID 25086187
- [Background] Regueiro M, Schraut W, Baidoo L, Kip KE, Sepulveda AR, Pesci M, Harrison J, Plevy SE. Infliximab prevents Crohn's disease recurrence after ileal resection. Gastroenterology. 2009 Feb;136(2):441-50.e1; quiz 716. doi: 10.1053/j.gastro.2008.10.051. Epub 2008 Oct 31. PMID 19109962
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospitalized Patients Receiving Infliximab: Patients hospitalized and scheduled to receive clinically indicated infliximab due to flare of moderate to severe UC.
Period: Overall Study
Arm/Group | Hospitalized Patients Receiving Infliximab
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hospitalized Patients Receiving Infliximab
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 34 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to be Colectomy Free at 3 Months
Description: Total number of participants to be colectomy free at 3 months
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients Receiving Infliximab
Number analyzed (Participants) | 13
Participants | 6

2. Primary Outcome: Number of Participants With the Need for Colectomy Assessed by Biomarker Levels
Description: Biomarkers markers ESR, CRP, TNF levels, and hemoglobin will be collected to assess relationships between colectomy an other potential biomarkers
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients Receiving Infliximab
Number analyzed (Participants) | 13
Participants | 13

3. Secondary Outcome: Number of Participants to be Colectomy Free at 1 Month
Description: Total number of participants to be colectomy free at 1 month
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Patients Receiving Infliximab
Number analyzed (Participants) | 13
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 3 months on all participants.
Arm/Group | Hospitalized Patients Receiving Infliximab
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02438410/Prot_000.pdf